CLINICAL TRIAL: NCT02582996
Title: National, Phase III, Multicenter, Randomized, Open, Parallel, to Evaluate the Efficacy, Safety and Superiority of Cefalium® Compared to the Tylenol® in the Treatment of Migraine Attacks
Brief Title: Cefalium® Compared to Tylenol® in the Treatment of Migraine Attacks
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic reasons of the company
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACH-CFL-03(01/14)
Record Dates: First submitted 2015-03-31; First posted 2015-10-21 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Migraine
Keywords: Headache; Aura; Migraine; Moderate to Severe
MeSH Terms: conditions — Migraine Disorders; Headache; Epilepsy | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cefalium® (Experimental): Acetaminophen+Caffeine+Dihydroergotamine+Metoclopramide.
  Interventions: Drug: Acetaminophen+Caffeine+Dihydroergotamine+Metoclopramide.
- Tylenol® (Active Comparator): Acetaminophen
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen+Caffeine+Dihydroergotamine+Metoclopramide. — The subject must manage 02 tablets of Cefalium right after a moderate to severe migraine.
  Other Names: Cefalium
  Arms: Cefalium®
Drug: Acetaminophen — The subject must manage 02 tablets of Tylenol right after a moderate to severe migraine.
  Other Names: Tylenol
  Arms: Tylenol®

SUMMARY:
National clinical trials, phase III, randomized, open, parallel, study of superiority, in which three hundred thirty-six (336) participants of both sexes, aged between 18 and 65 years will be randomly allocated to one of two treatment groups. The Group 01 will use Cefalium® and group 02 will use Tylenol®.

DETAILED DESCRIPTION:
Cefalium® is a combination of Caffeine + Paracetamol + dihydroergotamine mesylate + metoclopramide hydrochloride. The dihydroergotamine mesylate interacts with the serotonergic, dopaminergic and noradrenergic receptors, but it's mechanism is not totally known. The caffeine presents mechanisms that are not totally clear, but it may relieves the pain by activating of the central noradenosine pathway (pain suppressing system). The Metoclopramide hydrochloride presents an anti-emetic action and prokinetic action in the gastrointestinal tract.One of its properties is the inhibition of nausea and vomiting triggered by drugs such as ergotamine.Paracetamol, also called acetaminophen is an effective agent analgesic and antipyretic with weak anti-inflammatory activity.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both gender;
* Age older or equal to 18 and younger than 66 years if they have symptoms of migraine headache before 50 years of age;
* Presence of migraine headache with or without aura symptoms, at least 03 months prior to the study, the criteria defined by International Classification of Headache Disorders(ICHD)-II, 2004 (IHS International Headache Society) - Annex I;
* Subjects which are experiencing 2-6 migraine attacks per month with mild to moderate pain intensity in the last 3 months prior to screening visit;
* Participants which are able to distinguish migraine attacks to any other type of headache;
* Ability to understand and consent to participate in this clinical research, expressed by signing the Informed Consent Form (ICF).

Exclusion Criteria:

* Any clinical finding (clinical evaluation / physical) that is interpreted by the Investigator as a risk to the subject in the clinical trial;
* Subjects which had recent episodes of headache, with frequency equal or higher than 15 daily episodes per month, 3 months prior to the screening visit;
* Subjects with headache history defined by the ICHD-II criteria, 2004 IHS (International Headache Society) rated as:

  * Typical aura with non-migraine headache;
  * Typical aura without headache;
  * Familial Hemiplegic Migraine (FHM);
  * Sporadic Hemiplegic Migraine;
  * Basilar type Migraine;
* Any laboratorial finding that the Investigator consider a risk to subject of the study;
* Hypersensitivity to the drug components used during the study;
* Women in pregnancy or nursing period;
* Women in reproductive age who do not agree to use contraception acceptable [oral contraceptives, injectable contraceptives, intrauterine device (IUD), hormonal implants, barrier methods, hormonal patch and tubal ligation]; other than surgically sterile (bilateral oophorectomy or hysterectomy), postmenopausal for at least one (01) years or sexual abstinence;
* Inability to understand and answer to the functional categorical scale of the study, diary of symptoms, and not having accompanying to assist him/her;
* History of abuse, according to the principal investigator, of the alcohol, opioids, barbiturates, benzodiazepines and illicit drugs in the last 02 years, or abuse of drugs for headache including ergotamines or narcotics in the last 03 months;
* Subjects with prolonged hypotension, shock, sepsis, pheochromocytoma, hemorrhage, mechanical obstruction or perforation of the gastrointestinal tract
* Participants with glucose-6-phosphate dehydrogenase(G6PD) deficiency due to increased risk of hemolysis associated with the use of paracetamol;
* Subjects with history of epilepsy or presence of psychiatric illness of any kind, in the opinion of the investigator, that may interfere with adherence to treatment;
* Subjects with a malignant disease less than five years, or for more than five years, but without documentation about the remission/cure. As example: melanoma, leukemia, lymphoma, myeloproliferative diseases and renal cell carcinoma of any length should be excluded. Exceptions: Participants with basal cell skin cancers, squamous cell, and cervical cancer in situ may be eligible;
* Subjects which uses a preventive treatment and changed the dose in the last 02 weeks before the screening visit (V0);
* Subjects with hepatic or renal failure;
* Subjects that has participated in clinical trial protocols in the last twelve (12) months (National Board of Health- Resolution 251 of 07 August 1997, Part III, sub-item J), unless the investigator considers that there may be a direct benefit to it;
* Subjects who are in prohibited medication as described in item 10.2 of the Protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2020-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Pain relief of Cefalium® compared to Tylenol® | 2 hours
  Relief of pain 2 hours after taking medication, being considered to reduce the intensity from strong(3) or moderate(2), at baseline, to mild(1) or absent(0) 2 hours after taking the medication, according to the functional and behavioral debilitating categorical scale without use of rescue medication as annotations the diary of symptoms

SECONDARY OUTCOMES:
Pain decrease after use of investigational product, without a rescue medication | Up to 4 hours
  Number of participants with pain decrease in 2 hours and 4 hours after the use of the investigational product,at the first migraine attack with mild or moderate pain, with remission defined as no pain (0) in categorical scale debilitating functional and behavioral (4 point-scale), without use of a rescue medication
Pain decrease after use of the investigational product, without a rescue medication | 4 hours
  Number of participants with pain relief in 4 hours after the use of the investigational product, in the first migraine attack with mild or moderate pain,and is considered the relief reduction of at least 01 point in pain intensity from baseline, according to functional and behavioral debilitating categorical scale without use of a rescue medication;
Pain relief maintenance during the period 4-24 hours after use of investigational product | Up to 24 hours
  The maintenance will be observed if the relief reached the first 4 hours will remain at 24 hours after use of the investigational product, according to functional and behavioral debilitating categorical scale (4 point scale) without use of rescue medication during this period;
Nausea/vomiting Symptoms Free | Up to 4 hours
  Participants free of nausea/vomiting symptoms 2 and 4 hours after use of investigational product,at the first migraine attack of moderate to severe pain intensity, defined as the proportion of subjects with no symptoms of both among the participants have at least one symptom at baseline of migraine without use of a rescue medication during this period.
Photophobia/Phonophobia Symptoms Free | Up to 4 hours
  Participants free of photophobia/phonophobia symptoms 2 and 4 hours after use of investigational product, at the first migraine attack of moderate to severe pain intensity, defined as the proportion of subjects with no symptoms of both among the participants have at least one symptom at baseline of migraine without use of a rescue medication during this period.
Need of a rescue medication | Up to 24 hours
  Number of participants who use at least once the rescue medication in a 2-24 hours period after use of the investigational product.

OTHER OUTCOMES:
Variation in laboratory exams ratings | From baseline visit until 30 days after the end of the treatment
  Number of participants with any relevant variation in laboratory exams from baseline visit until 30 days after the end of the treatment
Variation in clinical exams ratings | From baseline visit until 30 days after the end of the treatment
  Number of participants with any relevant variation in clinical exams from baseline visit until 30 days after the end of the treatment
Variation in physical exams ratings | From baseline visit until 30 days after the end of the treatment
  Number of participants with any relevant variation in physical exams from baseline visit until 30 days after the end of the treatment
Participants with adverse events | From baseline visit until 30 days after the end of the treatment
  Number of participants with any adverse events from baseline visit until 30 days after the end of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thais Villa, Principal Investigator — Federal University of São Paulo
Locations (6):
- Brazil (6):
  - Centro de Pesquisa Clínica - CPEC / Associação Obras Sociais Irmã Dulce, Salvador, Estado de Bahia
  - Centro de Pesquisa Clínica Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Centro de Desenvolvimento em Estudos Clínicos Brasil - CDEC Brasil, São Paulo
  - Cepic - Centro Paulista de Investigação Clínica, São Paulo
  - CPCLIN - Centro de Pesquisas Clinicas Ltda, São Paulo
  - Universidade Federal de São Paulo - Núcleo de Gestão de Pesquisa/HU/FAP, São Paulo